CLINICAL TRIAL: NCT00979745
Title: A Phase III, Multicentre, Double-Blind, Randomised, Placebo-Controlled Study to Confirm the Safety and Efficacy of Subcutaneous Bioresorbable Afamelanotide Implants in Patients With Erythropoietic Protoporphyria (EPP)
Brief Title: Phase III Confirmatory Study in Erythropoietic Protoporphyria (EPP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CUV029
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Erythropoietic Protoporphyria
Keywords: Erythropoietic Protoporphyria; EPP; Afamelanotide
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — afamelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Afamelanotide (Experimental)
  Interventions: Drug: Afamelanotide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afamelanotide — One 16mg subcutaneous implant every 2 months for 9 months.
  Other Names: CUV1647
  Arms: Afamelanotide
Drug: Placebo — One 16mg subcutaneous implant every 2 months for 9 months.
  Arms: Placebo

SUMMARY:
Afamelanotide is a man-made drug being studied for use as a preventative medication for EPP sufferers. It is a synthetically produced analogue of human alpha melanocyte stimulating hormone (alpha-MSH) and is not yet available on the market.

The purpose of this study is to look at whether afamelanotide can reduce the number and severity of EPP symptoms when patients are exposed to light. This study will also look at how the drug is tolerated when taken by people with EPP.

The study will involve the use of an implant, which comes in the form of a small rod (approximately 2 cm x 0.15 cm) to be administered under the skin. The implant may contain the study drug afamelanotide or a placebo (inactive medication).

Over 450 subjects have been treated with afamelanotide to date with no serious safety concerns identified. For this study, afamelanotide has been formulated as a controlled release depot injection (implant). This means that the afamelanotide will be released slowly into the body over a few days. Once inserted, the implant will remain in the body after afamelanotide has been released and will slowly dissolve.

This study will help to provide more information about afamelanotide. This information will be used to determine the safety and efficacy (the ability of the drug to produce an effect) of this drug in EPP sufferers.

Up to 70 people will participate in this study from study sites across Europe.

DETAILED DESCRIPTION:
PURPOSE:

To determine whether afamelanotide can reduce the severity of phototoxic reactions in patients with EPP.

THEORETICAL FRAMEWORK:

EPP is a genetic photosensitivity disorder where the mainstays of management are covering up from sunlight, systemic beta carotene and the use of controlled courses of UVR treatment. One of the mechanisms for the protective effects of UVR treatment is the increase in melanin content of the skin. UVR treatment causes DNA damage to skin cells and increases the risk for skin cancers, hence it is unwise for this to be used on a recurring basis. Afamelanotide, through its ability to stimulate melanin production without causing the DNA damage associated with UVR treatment, appears to be a promising agent to combat this distressing disorder.

STUDY DESIGN:

This is a phase III, randomised, placebo controlled study to evaluate the safety and efficacy of subcutaneous implants of afamelanotide in patients suffering from EPP. The study will be performed in compliance with Good Clinical Practice (GCP) including the archiving of essential documents.

METHODOLOGY:

The target population consists of male and female participants. Up to 70 patients with diagnosed EPP (from past case history) and fulfilling the necessary inclusion/exclusion criteria will be enrolled. Potential study patients will be identified from each centre's records of patients with well characterised history (or documented diagnosis) of EPP.

Patients will be enrolled and will receive afamelanotide (16 mg implants) or placebo according to the following dosing regime:

* Group A will be administered active implants on Days 0, 60, 120, 180 and 240.
* Group B will be administered placebo implants on Days 0, 60, 120, 180 and 240.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a diagnosis of EPP (confirmed by elevated free protoporphyrin in peripheral erythrocytes) of sufficient severity that they have requested treatment to alleviate their symptoms.
* Aged 18 - 70 years (inclusive)
* Written informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* Any allergy to afamelanotide or the polymer contained in the implant or to lignocaine or other local anaesthetic to be used during the administration of study medication.
* EPP patients with significant hepatic involvement.
* Personal history of melanoma or dysplastic nevus syndrome.
* Current Bowen's disease, basal cell carcinoma, squamous cell carcinoma, or other malignant or premalignant skin lesions.
* Any other photodermatosis such as PLE, DLE or solar urticaria.
* Any evidence of clinically significant organ dysfunction or any clinically significant deviation from normal in the clinical or laboratory determinations.
* Acute history of drug or alcohol abuse (in the last 12 months).
* Patient assessed as not suitable for the study in the opinion of the Investigator (e.g. noncompliance history, allergic to local anaesthetics, faints when given injections or giving blood).
* Female who is pregnant (confirmed by positive serum β-HCG pregnancy test prior to baseline) or lactating.
* Females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device).
* Sexually active men with partners of child bearing potential not using barrier contraception during the trial and for a period of three months thereafter.
* Participation in a clinical trial of an investigational agent within 30 days prior to the screening visit.
* Prior and concomitant therapy with medications which may interfere with the objectives of the study, including drugs that cause photosensitivity or skin pigmentation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Anstey, MBBS, FRCP, Principal Investigator — St Woolos Hospital, Newport; Jorge Frank, MD, PhD, Principal Investigator — Academisch Ziekenhuis Maastricht; Raili Kauppinen, MD, PhD, Principal Investigator — University Central Hospital of Helsinki; Eric JG Sijbrands, MD, PhD, Principal Investigator — Erasmus Medical Center; Jean-Charles Deybach, MD. PhD, Principal Investigator — Centre Francais des Porphyries, Hopital Louis Mourier, Colombes, France; Sandra Hanneken, MD, Principal Investigator — Heinrich-Heine Universität, Düsseldorf, Germany; Gillian M Murphy, MD PhD, Principal Investigator — Beaumont Hospital, Dublin, Ireland; Lesley E Rhodes, MD PhD, Principal Investigator — Hope Hospital, University of Manchester, UK
Locations (8):
- HUS:n Iho-ja allergiasairaala (Skin and Allergy Hospital), Helsinki, Finland
- Centre Français des Porphyries, Hôpital Louis Mourier, Colombes, Cedex, France
- Department of Dermatology , Heinrich-Heine-University Duesseldorf, Düsseldorf, Germany
- Beaumont Hospital, Department of Dermatology, Dublin, Ireland
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Erasmus Medical Center, Rotterdam
- United Kingdom (2):
  - St Woolos Hospital, Newport, Wales
  - Photobiology Unit - Hope Hospital, University of Manchester, Manchester

REFERENCES:
- [Derived] Langendonk JG, Balwani M, Anderson KE, Bonkovsky HL, Anstey AV, Bissell DM, Bloomer J, Edwards C, Neumann NJ, Parker C, Phillips JD, Lim HW, Hamzavi I, Deybach JC, Kauppinen R, Rhodes LE, Frank J, Murphy GM, Karstens FPJ, Sijbrands EJG, de Rooij FWM, Lebwohl M, Naik H, Goding CR, Wilson JHP, Desnick RJ. Afamelanotide for Erythropoietic Protoporphyria. N Engl J Med. 2015 Jul 2;373(1):48-59. doi: 10.1056/NEJMoa1411481. PMID 26132941

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Afamelanotide: administered afamelanotide implants on Days 0, 60, 120, 180 and 240.
- Placebo: administered placebo implants on Days 0, 60, 120, 180 and 240.
Period: Overall Study
Arm/Group | Experimental: Afamelanotide | Placebo
Started | 38 | 36
Completed | 34 | 34
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Afamelanotide | Placebo | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (13) | 38.6 (11.6) | 38.45 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 17 | 20 | 37

OUTCOME MEASURES:

1. Primary Outcome: The Duration of Direct Sunlight Exposure Between 10:00 and 15:00 Hours on Days When Patients Did Not Report Phototoxicity-related Pain (Likert Pain Scale Score of 0)
Time Frame: From baseline to Day 270
Measure: Median (Full Range); unit: Hours
Arm/Group | Experimental: Afamelanotide | Placebo
Number analyzed (Participants) | 38 | 36
Hours | 6.0 [0 to 192.5] | 0.75 [0 to 34.8]

2. Secondary Outcome: Number of Phototoxic Reactions
Time Frame: 9 months
Reporting Status: Not Posted

3. Secondary Outcome: Quality of Life Measured by Patient Completed Questionnaire
Time Frame: 9 months
Reporting Status: Not Posted

4. Secondary Outcome: Free Protoporphyrin IX Level
Time Frame: 9 months
Reporting Status: Not Posted

5. Secondary Outcome: Treatment Emergent Adverse Events
Time Frame: 9 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Experimental: Afamelanotide: Afamelanotide implants administered on Days 0, 60, 120, 180 and 240.
- Placebo: Placebo implants administered on Days 0, 60, 120, 180 and 240.
Arm/Group | Experimental: Afamelanotide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 16/38 | 12/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Afamelanotide (N=38) | Placebo (N=36)
Implant site discolouration (General disorders) | 4 | 0
Blood urine present (Investigations) | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 6 | 3
Dizziness (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No